CLINICAL TRIAL: NCT07107672
Title: Mass Balance and Biotransformation Study of [14C]X842 in Healthy Adult Male Subjects in China
Brief Title: Mass Balance Study of [14C]X842 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Sinorda Biomedicine Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SND-X842-102
Record Dates: First submitted 2025-07-14; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Reflux Esophagitis; X842; Pharmacokinetics, PK; [14C]X842; linaprazan
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis, Peptic

STUDY DESIGN:
Intervention Model Description: The study plans to enroll 6 to 8 healthy male subjects in China to ensure at least 4 evaluable subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]X842 suspension approximately 50 mg/ 100 µCi[14C]X842 (Experimental): a single oral administration of approximately 50 mg/ 100 µCi [14C]X842 suspension orally on an empty stomach on day 1
  Interventions: Drug: [14C]X842

INTERVENTIONS:
Drug: [14C]X842 — 50 mg/100 µCi [14C] X842 suspension
  Other Names: [14C]X842 suspension

SUMMARY:
This study is a single-site, single-dose, non-randomized, open-label study to assess the absorption, metabolism, and excretion profile of [14C]X842 in healthy adult male subjects. The study plans to enroll 6 to 8 healthy male subjects in China to ensure at least 4 evaluable subjects.

DETAILED DESCRIPTION:
The healthy male subjects will be screened no more than 14 days before the dose (D-14 through D-3) and admitted to the clinical research center 2 days before the dose (D-2). The subjects will receive a single oral administration of approximately 50 mg/100 µCi [14C]X842 suspension orally on an empty stomach on day 1.

Urine and feces samples will be all collected from the subjects before and at specified intervals between 0 and 312 hours after taking the drug and blood samples will be collected at specified time points between 0 and 216 hours before and after taking the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males;
2. Age: 18 to 45 years (inclusive)
3. Body weight: ≥50 kg with body mass index (BMI) between 19.0 and 26.0 kg/m² (inclusive);
4. Fully understand the trial objectives, requirements, procedures, and potential adverse reactions; voluntarily participate; able to complete the study per protocol and comply with regulations; informed consent obtained in compliance with GCP;
5. The subjects were able to communicate well with the researchers and complete the trial in accordance with the provisions of the protocol.

Exclusion Criteria:

- Auxiliary Examinations:

1. Subjects with abnormal and clinically significant findings in Physical examination, Vital signs, Laboratory tests (including hematology, blood biochemistry, coagulation, urinalysis, fecal occult blood),Thyroid function, 12-lead ECG, Anteroposterior chest X-ray, Abdominal ultrasound, and/or other clinically relevant investigations;
2. Subjects testing positive for: Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV-Ab), Human immunodeficiency virus antibody (HIV-Ab),Treponema pallidum antibody (syphilis screening);

   -Medication History:
3. Subjects with use of any medications known to inhibit or induce hepatic drug-metabolizing enzymes within 30 days prior to screening；
4. Subjects with use of any prescription medications, over-the-counter drugs, Chinese herbal medicines, or dietary supplements (e.g., vitamins, calcium) within 14 days prior to screening;

   -Disease and Surgical History
5. History of any clinically significant disease or condition that the investigator deems may affect the trial results, including but not limited to diseases of the circulatory, respiratory, endocrine, nervous, digestive, urinary systems, or blood, immune, psychiatric, and metabolic disorders;
6. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade de pointes, ventricular tachycardia, atrioventricular block, long QT syndrome, or family history thereof (as evidenced by genetic confirmation or sudden cardiac death of close relatives at a young age);
7. Major surgery within 6 months prior to screening, or incompletely healed surgical wounds; Major surgery includes, but is not limited to, any procedure with significant bleeding risk, prolonged general anesthesia, open biopsy, or significant traumatic injury;
8. Subjects have prone to allergies, such as a known history of hypersensitivity to two or more substances; or individuals deemed by the investigator as potentially allergic to the trial drug or its excipients;
9. Subjects with regular/ongoing hematochezia, irritable bowel syndrome, inflammatory bowel disease;

   -life style
10. Subjects with habitual constipation or diarrhea;
11. Subjects who has the history of alcoholism or regular alcohol consumption within 6 months prior to screening, defined as consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine), and inability to abstain during the trial period; or a breath alcohol test result ≥ 0 mg/dL at screening;
12. Subjects who have smoked more than 5 cigarettes per day or habitually using nicotine-containing products within 3 months prior to screening, or who are unable to stop using any tobacco products during the trial;
13. Subjects who have a history of drug abuse within three months prior to the screening period or whose urine test for prohibited drugs (morphine, methamphetamine, ketamine, dimethylene dioxyethanol, tetrahydrocannabinic acid) is positive during the screening;
14. Subjects who has habitually consumption of grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages and are unable to quit during the trial period;
15. Subjects who are exposed to radioactive work conditions for a long time, or have significant radiation exposure (≥ 2 chest/abdominal CTs, or ≥ 3 other types of X-ray examinations) within 1 year before the first dose, or have participated in a radiopharmaceutical labeled trial;
16. Subjects with a history of blood or needle phobia, and those who have difficulty in blood collection or cannot tolerate venipuncture blood collection;
17. Subjects have participated in any other clinical trial (including trials of investigational drugs or medical devices, etc.) within 3 months prior to the screening period.
18. Subjects who have received any vaccination within 1 month prior to screening or plan to receive any vaccination during the study period;
19. subjects who plan to conceive or donate sperm during the trial period or within 1 year after trial completion, or those who do not agree that the subject and their partner must use highly effective contraception during the trial period and for 1 year after trial completion;
20. Subjects who have lost blood or donated blood (200mL), or received blood transfusions within 3 month before the screening period.
21. Subjects who are unsuitable for the study participation for other reasons at the discretion of the investigator;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Mass balance: the cumulative excretion rate | 22 days
  To collect the total radioactive substances in excreta (urine and feces) and to calculate the cumulative excretion rate
Tmax (time to maximum observed concentration) | 22 days
  Tmax parameters of the total radioactivity in plasma
Cmax(maximum concentration) | 22 days
  Cmax parameters of the total radioactivity in plasma
AUC(area under curve) | 22 days
  AUC parameters of the total radioactivity in plasma
t1/2 (terminal elimination half-life) | 22 days
  t1/2 parameters of the total radioactivity in plasma
MRT (mean residence time) | 22 days
  MRT parameters of the total radioactivity in plasma
Vd/F(apparent volume of distribution) | 22 days
  Vd/F parameters of the total radioactivity in plasma
whole blood/plasma ratio for the total radioactivity concentration at different time points | 22 days
  whole blood/plasma ratio for the total radioactivity concentration at different time points
Percentage of the drug and its metabolites in plasma, urine and feces to the administered dose | 22 days
  Exposure in plasma; percentage of the drug and its metabolites in urine and feces to the administered dose; identification of major metabolites in plasma, urine and feces

SECONDARY OUTCOMES:
The nature and severity of AEs based on NCI-CTC AE V5.0 | 22 days
  The nature and severity of adverse events were adjudicated in accordance with the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0)
The nature and incidence and severity of SAEs based on NCI-CTC AE V5.0 | 22 days
  The nature and severity of serious adverse events were adjudicated in accordance with the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0)
12-Electrocardiograms (ECG) | 22 days
  the data collection of heart rate, PR interval, QRS interval, QT, QTc, on D-1 and 2 hours (±30 min) after administration
vital signs of pulse | 22 days
  pulse (beats per minute)
vital signs of body temperature | 22 days
  body temperature (℃)
vital signs of blood pressure | 22 days
  measurements included systolic (mmHg) and diastolic (mmHg).
vital signs of respiratory rate | 22 days
  respiratory rate (breaths per minute).
Hematology - Number of participants with clinically significant abnormalities | 22 days
  including White blood cell count, lymphocyte count, neutrophil count, red blood cell count, hemoglobin, platelet count
Blood Chemistry - Number of participants with clinically significant abnormalities | 22 days
  Blood Biochemistry including: Total Bilirubin (TBIL), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma-Glutamyl Transferase (GGT), Alkaline Phosphatase (ALP), Total Protein (TP), Albumin (ALB), Urea, Creatinine (Cr), Uric Acid (UA), Glucose (GLU), Total Cholesterol (TC), High-Density Lipoprotein Cholesterol (HDL-C), Low-Density Lipoprotein Cholesterol (LDL-C), Triglycerides (TG), Potassium (K+), Sodium (Na+), Chloride (Cl-), Lactate Dehydrogenase (LDH), Creatine Kinase (CK), Amylase (AMY).
Coagulation - Number of participants with clinically significant abnormalities | 22 days
  including Prothrombin Time (PT), Thrombin Time (TT), Activated Partial ,, hromboplastin Time (APTT/aPTT)，Fibrinogen (FIB/Fg), International Normalized Ratio (INR)
Urinalysis - Number of participants with clinically significant abnormalities | 22 days
  Urinalysis including Urinary protein, urine sugar, urine ketone bodies, red blood cells, white blood cells, pH value
Fecal Occult Blood Test (FOBT) - Number of participants with positive result | 22 days
  Fecal Occult Blood Test (FOBT) result

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China